"Young Adult EC Use and Respiratory Outcomes (K01)"

Power Analyses. For Aims 1 and 2: The use of repeated measures and longitudinal methodology allow for greater detection of moderate effect sizes associated with decreased in markers of respiratory health, increases in nicotine addiction, changes in EC and/or OTP use patterns, and frequency/quantity of EC use. For each repeated measures analysis of variance (ANOVA) and multivariate analysis of variance (MANOVA) we are 95% powered to find moderate effect sizes. For Aim 3: Power was calculated using MPlus Monte Carlo estimation informed by published and preliminary studies. To test power for MLM, we first examined power with Optimal Design using repeated measures. We then repeated our power analyses in MPlus Monte Carlo estimation, building on published MLM simulations and using 1000 replications to confirm stability of each model, to better capture the complexity of the separate models, including cross-level interactions. For the EMA analyses, the power of the statistical test depends on the total effective sample size (ESS) and the statistical model used. The total ESS is the number of statistically independent observations available for this study. The number of statistically independent observations is the total number of observations (number of participants x number of data collections) adjusted for within-individual correlations. As the within-individual, or intra-class, correlation (ICC) increases, the ESS decreases. The following formula illustrates this relationship, whereby the effective sample size is equal to nm/(1+(m-1)p), where n = number of participants; m = number of repeated measures foreach participant; and  $\rho = ICC.94$  In sum, even assuming effects as small as .10 (well below expected effect), we will be well powered (> .85) to identify effects across analyses.

<u>Data Analytic Overview.</u> Analyses will be conducted using SAS, R and MPlus. <u>For Aims 1 and 2</u>, distribution plots will be carried out on all data to assess for normality, and any non-Gaussian data were evaluated with either Wilcoxon signed rank test or, where appropriate, data will be logarithmically transformed before analysis. Comparisons of continuous data will be made by an overall analysis of variance, followed by Bonferroni corrected, multiple-range testing, to obviate multiple pairwise comparisons, with the overall α error set at .05 (2tailed). <u>For Aim 3</u>, as appropriate, alternate estimators to address expected and observed characteristics (e.g., Poisson distribution, zero-inflation) will be used. MPlus permits frequentist and Bayesian estimation for models with missing data. Bayesian procedures allow multiple imputation of multiple datasets subsequently used with parameter estimates averaged across imputed datasets. Multiple imputation will virtually always outperform older methods of managing missing data (e.g., listwise deletion) with regard to both accuracy and power, making it the preferred approach. <sup>72, 73</sup> Measurement models will be formally tested. If analyses do not support the presence of the expected unitary constructs, subsequent analyses will examine aims as defined by observed variables. Model invariance tests will also be used to assess appropriate statistical treatment of gender; if measurement invariance is not observed, analyses will be stratified by gender.

<u>Aim 1: Hypotheses 1a and 1b:</u> We will use two-way repeated measures ANOVA and MANOVA with Tukey adjustment to examine differences between the measures of respiratory health (pulmonary functioning, NELF samples) and EMA data (five two-week monitoring periods). For <u>H1a</u>, two-way repeated measures ANOVA will compare mean differences between pulmonary and respiratory markers and user status (EC-exclusive vs. neverusers). For <u>H1b</u>, we will use MANOVA models to examine changes in frequency/quantity of EC use and nicotine dependence (significant increases in HONC scores) across each session with respiratory and pulmonary functioning.

<u>Aim 2 Hypotheses 2a and 2b:</u> We will use two-way repeated measures analysis of variance and multivariate analysis of variance with Tukey-adjustment to examine differences between the number of vape sessions per day and time spent vaping with pulmonary functioning across each EMA monitoring period. For <u>H2a</u>, two-way repeated measures ANOVA will compare mean differences between pulmonary and frequency/quantity of EC use. For <u>H2b</u>, we use MANOVA models to examine changes in pulmonary functioning and the experimentation of OTP in conjunction with EC-use across the 1-year monitoring period.

Exploratory Aim 3: Hypotheses H3a: We will use multilevel models (MLM) to examine the daily-level associations between the frequency/quantity of EC use experimentation and pulmonary functioning. These models will allow us to examine the within-person associations between EC use and pulmonary functioning, using Curran and Baurer's<sup>95</sup> procedures for disaggregating within-person and between-person effects using two level analysis in multilevel modeling. These models will also allow for the examination of cross-level interactions among between and within-person factors. Specifically, we will be able to examine the role of daily within-person fluctuations in

frequency/quantity of EC use in its links to pulmonary functioning. Further, we will be able to assess the potential differences by user status as well as baseline respiratory health. Significant interactions will be probed using Preacher, Curran, & Bauer's 6 computational tools.

## **Bibliography**

- 1. Pai AL, Tackett A, Ittenbach RF, Goebel J. Psychosocial Assessment Tool 2.0 \_General: validity of a psychosocial risk screener in a pediatric kidney transplant sample. *Pediatric transplantation*. 2012;16(1):92-98.
- 2. Pai AL, Rausch J, Tackett A, Marsolo K, Drotar D, Goebel J. System for integrated adherence monitoring: Real-time non-adherence risk assessment in pediatric kidney transplantation. *Pediatric transplantation*. 2012;16(4):329-334.
- 3. Pai AL, Tackett A, Hente EA, Ernst MM, Denson LA, Hommel KA. Assessing psychosocial risk in pediatric inflammatory bowel disease: validation of the Psychosocial Assessment Tool 2.0 \_General. *Journal of pediatric gastroenterology and nutrition.* 2014;58(1).
- 4. Tackett AP, Peugh JL, Wu YP, Pai AL. Parent Medication Barriers Scale (PMBS): A preliminary investigation of factor structures with hematopoietic stem cell transplant recipients. *Children's Health Care*. 2016;45(2):177-191.
- 5. Tackett AP L, W.V., Meier, E, Suorsa, K.I, Wagener, T.L, & Mullins, L.L. Tobacco usestatus as a function of health care utilization attitudes/beliefs. The Association for Behavioral and Cognitive Therapies; 2013; Nashville, TN.
- 6. Tackett AP, Leavens EL, Wiedenmann A, et al. Preliminary exploration of secondhand smoke exposure in youth with Sickle Cell Disease: biochemical verification, pulmonary functioning, and health care utilization. *Psychology, health & medicine.* 2018:1-8.
- 7. Turner E, Fedele DA, Thompson L, Salloum RG. Patterns of electronic cigarette use in youth with asthma: Results from a nationally representative sample. *Annals of Allergy, Asthma & Immunology.* 2018;120(2):220-222.
- 8. Reid KM, Forrest JR, Porter L. Tobacco Product Use Among Youths With and Without Lifetime Asthma—Florida, 2016. *Morbidity and Mortality Weekly Report*. 2018;67(21):599.
- 9. Choi K, Bernat D. E-cigarette use among Florida youth with and without asthma. *American journal of preventive medicine*. 2016;51(4):446-453.
- 10. Schweitzer RJ, Wills TA, Tam E, Pagano I, Choi K. E-cigarette use and asthma in a multiethnic sample of adolescents. *Preventive medicine*. 2017;105:226-231.
- 11. Tackett, A.P., Keller-Hamilton, B., Hébert, E.T., Smith, C.E., Metcalf, J., Queimado, L., Stevens, E.M., Wallace, S., McQuaid, E.L. & Wagener, T.L. (in press). Associations of Respiratory Symptoms among Youth E-Cigarette Users: Results from the PATH Study. JAMA Network Open.
- 12. Roberts CM, Tackett, A.P. Leavens, E.L.S., Edwards, C., Stevens, E.M., Hébert, E.L., Villanti, PhD, A.C., Pearson, J.L., & Wagener, T.L. . JUUL Perceived Drug Effects and Preferences between Emerging Adults, Young Adults, and Older Adults. under review.
- 13. Tackett A, Edwards, C, Roberts, CM, Stevens, E, Leavens, ELS, and Wagener, TL. Examining Other Tobacco and Marijuana Use Among Experimenters and Current Users of JUUL. under review.
- 14. Searby L, Ballenger J, Tripses J. Climbing the ladder, holding the ladder: The mentoring experiences of higher education female leaders. *Advancing Women in Leadership*. 2015;35:98-107.
- 15. United States Department of Health and Human Services. The health consequences of smoking—50 years of progress: a report of the Surgeon General. *Atlanta, GA: US Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Office on Smoking and Health.* 2014;17.
- 16. United Stated Department of Health and Human Services. A Report of the Surgeon General; US Department of Health and Human Services, Centers for Disease Control and Prevention. *National Center for Chronic Disease Prevention and Health Promotion, Office on Smoking and Health: Atlanta, GA, USA.* 2016.
- 17. Carpenter CM, Wayne GF, Pauly JL, Koh HK, Connolly GN. New cigarette brands with flavors that appeal to youth: tobacco marketing strategies. *Health Affairs*. 2005;24(6):1601-1610.
- 18. Gostin LO, Glasner AY. E-cigarettes, vaping, and youth. *Jama*. 2014;312(6):595-596.
- 19. Lempert LK, Glantz S. Packaging colour research by tobacco companies: the pack as a product characteristic. *Tobacco control.* 2017;26(3):307-315.

- 20. Zhu S-H, Sun JY, Bonnevie E, et al. Four hundred and sixty brands of e-cigarettes and counting: implications for product regulation. *Tobacco control.* 2014;23(suppl 3):iii3-iii9.
- 21. Gibson-Young LM. JUULING: What kids don't know will hurt them. *Pediatrics*. 2018;35(6).
- 22. Goniewicz ML, Boykan R, Messina CR, Eliscu A, Tolentino J. High exposure to nicotine among adolescents who use Juul and other vape pod systems ('pods'). *Tobacco control*. 2018:tobaccocontrol2018-054565.
- 23. Huang J, Duan Z, Kwok J, et al. Vaping versus JUULing: how the extraordinary growth and marketing of JUUL transformed the US retail e-cigarette market. *Tobacco control*. 2018:tobaccocontrol-2018054382.
- 24. Willett JG, Bennett M, Hair EC, et al. Recognition, use and perceptions of JUUL among youth and young adults. *Tobacco control*. 2018:tobaccocontrol-2018-054273.
- 25. Kiljander T, Helin T, Venho K, Jaakkola A, Lehtimäki L. Prevalence of asthma–COPD overlap syndrome among primary care asthmatics with a smoking history: a cross-sectional study. *NPJ primary care respiratory medicine*. 2015;25:15047.
- 26. Usmani OS, Singh D, Spinola M, Bizzi A, Barnes PJ. The prevalence of small airways disease in adult asthma: a systematic literature review. *Respiratory medicine*. 2016;116:19-27.
- 27. Torres A, Blasi F, Dartois N, Akova M. Which individuals are at increased risk of pneumococcal disease and why? Impact of COPD, asthma, smoking, diabetes, and/or chronic heart disease on communityacquired pneumonia and invasive pneumococcal disease. *Thorax.* 2015:thoraxjnl-2015-206780.
- 28. Liu Y, Pleasants RA, Croft JB, et al. Smoking duration, respiratory symptoms, and COPD in adults aged≥ 45 years with a smoking history. *International journal of chronic obstructive pulmonary disease*. 2015;10:1409.
- 29. Dhariwal J, Tennant RC, Hansell DM, et al. Smoking cessation in COPD causes a transient improvement in spirometry and decreases micronodules on high-resolution CT imaging. *Chest.* 2014;145(5):1006-1015.
- 30. Leone FT, Carlsen K-H, Chooljian D, et al. Recommendations for the Appropriate Structure, Communication, and Investigation of Tobacco Harm Reduction Claims. An Official American Thoracic Society Policy Statement. *American journal of respiratory and critical care medicine*. 2018;198(8):e90e105.
- 31. Abram A, Zeller M. FDA's New Plan to Combat Tobacco's Staggering Public Health Toll. *Annals of the American Thoracic Society.* 2018(ja).
- 32. Tsai J, Walton K, Coleman BN, et al. Reasons for electronic cigarette use among middle and high school students—National Youth Tobacco Survey, United States, 2016. *Morbidity and Mortality Weekly Report*. 2018;67(6):196.
- 33. Leventhal AM, Strong DR, Kirkpatrick MG, et al. Association of electronic cigarette use with initiation of combustible tobacco product smoking in early adolescence. *Jama*. 2015;314(7):700-707.
- 34. Wang TW, Gentzke A, Sharapova S, Cullen KA, Ambrose BK, Jamal A. Tobacco Product Use Among Middle and High School Students—United States, 2011–2017. *Morbidity and Mortality Weekly Report.* 2018;67(22):629.
- 35. Truth Inititaive. Tobacco Rates in Oklahoma. 2018; <a href="https://truthinitiative.org/tobacco-use-oklahoma.">https://truthinitiative.org/tobacco-use-oklahoma.</a>
- 36. McGinley L. FDA chief calls youth e-cigarettes and 'epidemic'. *The Washington Post.* September 12, 2018, 2018.
- 37. Rohde JA, Noar SM, Horvitz C, Lazard AJ, Ross JC, Sutfin EL. The Role of Knowledge and Risk Beliefs in Adolescent E-Cigarette Use: A Pilot Study. *International journal of environmental research and public health.* 2018;15(4).
- 38. Soneji S, Barrington-Trimis JL, Wills TA, et al. Association between initial use of e-cigarettes and subsequent cigarette smoking among adolescents and young adults: a systematic review and metaanalysis. *JAMA pediatrics*. 2017;171(8):788-797.
- 39. Miech R, Patrick ME, O'malley PM, Johnston LD. E-cigarette use as a predictor of cigarette smoking: results from a 1-year follow-up of a national sample of 12th grade students. *Tobacco control*. 2017:tobaccocontrol-2016-053291.

- 40. Barrington-Trimis JL, Urman R, Berhane K, et al. E-cigarettes and future cigarette use. *Pediatrics*. 2016;138(1):e20160379.
- 41. Primack BA, Soneji S, Stoolmiller M, Fine MJ, Sargent JD. Progression to traditional cigarette smoking after electronic cigarette use among US adolescents and young adults. *JAMA pediatrics*. 2015;169(11):1018-1023.
- 42. Wills TA, Knight R, Sargent JD, Gibbons FX, Pagano I, Williams RJ. Longitudinal study of e-cigarette use and onset of cigarette smoking among high school students in Hawaii. *Tobacco control*. 2017;26(1):34-39.
- 43. Chassin L, Presson CC, Pitts SC, Sherman SJ. The natural history of cigarette smoking from adolescence to adulthood in a midwestern community sample: multiple trajectories and their psychosocial correlates. *Health Psychology*. 2000;19(3):223.
- 44. Hair E, Bennett M, Williams V, et al. Progression to established patterns of cigarette smoking among young adults. *Drug and alcohol dependence*. 2017;177:77-83.
- 45. Chen K, Kandel DB. The natural history of drug use from adolescence to the mid-thirties in a general population sample. *American journal of public health*. 1995;85(1):41-47.
- 46. Soneji S, Sargent J, Tanski S. Multiple tobacco product use among US adolescents and young adults. *Tobacco control.* 2016;25(2):174-180.
- 47. Bombard JM, Rock VJ, Pederson LL, Asman KJ. Monitoring polytobacco use among adolescents: do cigarette smokers use other forms of tobacco? *Nicotine & Tobacco Research*. 2008;10(11):1581-1589.
- 48. Cavazos-Rehg PA, Krauss MJ, Spitznagel EL, Grucza RA, Bierut LJ. Youth tobacco use type and associations with substance use disorders. *Addiction*. 2014;109(8):1371-1380.
- 49. Benowitz NL. Nicotine addiction. New England Journal of Medicine. 2010;362(24):2295-2303.
- 50. DiFranza JR, Savageau JA, Fletcher K, et al. Susceptibility to nicotine dependence: the Development and Assessment of Nicotine Dependence in Youth 2 study. *Pediatrics*. 2007;120(4):e974-e983.
- 51. Wheeler KC, Fletcher KE, Wellman RJ, Difranza JR. Screening adolescents for nicotine dependence: the Hooked On Nicotine Checklist. *Journal of Adolescent Health*. 2004;35(3):225-230.
- 52. Peirsman EJ, Carvelli TJ, Hage PY, et al. Exhaled nitric oxide in childhood allergic asthma management: a randomised controlled trial. *Pediatric pulmonology.* 2014;49(7):624-631.
- 53. Moradzadeh R, Mansournia MA, Baghfalaki T, Nadrian H, Gustafson P, McCandless LC. The impact of maternal smoking during pregnancy on childhood asthma: adjusted for exposure misclassification; results from the National Health and Nutrition Examination Survey, 2011–2012. *Annals of epidemiology.* 2018.
- 54. Jensen RP, Luo W, Pankow JF, Strongin RM, Peyton DH. Hidden formaldehyde in e-cigarette aerosols. 2015.
- 55. Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. *Therapeutic advances in drug safety.* 2014;5(2):67-86.
- 56. Callahan-Lyon P. Electronic cigarettes: human health effects. *Tobacco control.* 2014;23(suppl 2):ii36ii40.
- 57. Bishop E, Haswell L, Adamson J, Costigan S, Thorne D, Gaca M. An approach to testing undiluted ecigarette aerosol in vitro using 3D reconstituted human airway epithelium. *Toxicology in Vitro*. 2018.
- 58. Gerloff J, Sundar IK, Freter R, et al. Inflammatory response and barrier dysfunction by different ecigarette flavoring chemicals identified by gas chromatography–mass spectrometry in e-liquids and evapors on human lung epithelial cells and fibroblasts. *Applied in vitro toxicology.* 2017;3(1):28-40.
- 59. Allen JG, Flanigan SS, LeBlanc M, et al. Flavoring chemicals in e-cigarettes: diacetyl, 2, 3pentanedione, and acetoin in a sample of 51 products, including fruit-, candy-, and cocktail-flavored ecigarettes. *Environmental health perspectives*. 2015;124(6):733-739.
- 60. McConnell R, Barrington-Trimis JL, Wang K, et al. Electronic cigarette use and respiratory symptoms in adolescents. *American journal of respiratory and critical care medicine*. 2017;195(8):1043-1049.
- 61. Wang MP, Ho SY, Leung LT, Lam TH. Electronic cigarette use and respiratory symptoms in Chinese adolescents in Hong Kong. *JAMA pediatrics*. 2016;170(1):89-91.

- Ratajczak A, Feleszko W, Smith DM, Goniewicz M. How close are we to definitively identifying the respiratory health effects of e-cigarettes? *Expert review of respiratory medicine*. 2018(just-accepted). 63. Urman R, Barrington-Trimis J, Liu F, et al. Prospective Follow-Up of Respiratory Symptoms Among Young Adults with a History of Electronic Cigarette Use. In: *C16. Cigarette, E-cigarette, and Marijuana Smoking: Human and Mouse Studies*. American Thoracic Society; 2018:A4451-A4451.
- 64. Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Shortterm pulmonary effects of using an electronic cigarette: impact on respiratory flow resistance, impedance, and exhaled nitric oxide. *Chest.* 2012;141(6):1400-1406.
- 65. Chun LF, Moazed F, Calfee CS, Matthay MA, Gotts JE. Pulmonary toxicity of e-cigarettes. *American Journal of Physiology-Lung Cellular and Molecular Physiology*. 2017;313(2):L193-L206.
- 66. Kleinjan M, Engels RC, DiFranza JR. Parental smoke exposure and the development of nicotine craving in adolescent novice smokers: the roles of DRD2, DRD4, and OPRM1 genotypes. *BMC pulmonary medicine*. 2015;15(1):115.
- 67. Marini S, Buonanno G, Stabile L, Ficco G. Short-term effects of electronic and tobacco cigarettes on exhaled nitric oxide. *Toxicology and applied pharmacology.* 2014;278(1):9-15.
- 68. Dicpinigaitis PV, Chang AL, Dicpinigaitis AJ, Negassa A. Effect of e-cigarette use on cough reflex sensitivity. *Chest.* 2016;149(1):161-165.
- 69. Manigrasso M, Buonanno G, Fuoco FC, Stabile L, Avino P. Aerosol deposition doses in the human respiratory tree of electronic cigarette smokers. *Environmental Pollution*. 2015;196:257-267.
- 70. Fernández E, Ballbè M, Sureda X, Fu M, Saltó E, Martínez-Sánchez JM. Particulate matter from electronic cigarettes and conventional cigarettes: a systematic review and observational study. *Current environmental health reports.* 2015;2(4):423-429.
- 71. Farsalinos KE, Spyrou A, Tsimopoulou K, Stefopoulos C, Romagna G, Voudris V. Nicotine absorption from electronic cigarette use: comparison between first and new-generation devices. *Scientific reports*. 2014;4:4133.
- 72. Farsalinos KE, Spyrou A, Stefopoulos C, et al. Nicotine absorption from electronic cigarette use: comparison between experienced consumers (vapers) and naïve users (smokers). *Scientific reports*. 2015;5:11269.
- 73. Behar R, Davis B, Wang Y, Bahl V, Lin S, Talbot P. Identification of toxicants in cinnamon-flavored electronic cigarette refill fluids. *Toxicology in vitro*. 2014;28(2):198-208.
- 74. Robinson R, Hensel E, Morabito P, Roundtree K. Electronic cigarette topography in the natural environment. *PloS one*. 2015;10(6):e0129296.
- 75. Hammond D, Fong GT, Cummings KM, Hyland A. Smoking topography, brand switching, and nicotine delivery: results from an in vivo study. *Cancer Epidemiology and Prevention Biomarkers*. 2005;14(6):1370-1375.
- 76. Lerner CA, Sundar IK, Yao H, et al. Vapors produced by electronic cigarettes and e-juices with flavorings induce toxicity, oxidative stress, and inflammatory response in lung epithelial cells and in mouse lung. *PloS one*. 2015;10(2):e0116732.
- 77. Gass JC, Germeroth LJ, Wray JM, Tiffany ST. The reliability and stability of puff topography variables in non-daily smokers assessed in the laboratory. *Nicotine & Tobacco Research*. 2015;18(4):484-490.
- 78. Salepci B, Caglayan B, Fidan A, et al. The effect of pulmonary function testing on the success of smoking cessation. *Respiratory care*. 2016:respcare. 04490.
- 79. Barrington-Trimis JL, Urman R, Leventhal AM, et al. E-cigarettes, cigarettes, and the prevalence of adolescent tobacco use. *Pediatrics*. 2016:e20153983.
- 80. Gilreath TD, Leventhal A, Barrington-Trimis JL, et al. Patterns of alternative tobacco product use: emergence of hookah and e-cigarettes as preferred products amongst youth. *Journal of Adolescent Health*. 2016;58(2):181-185.
- 81. Pew Research Center. Teens, Social Media & Technology 2018. 2018; http://www.pewinternet.org/2018/05/31/teens-social-media-technology-2018/
- 82. Watkins SL, Glantz SA, Chaffee BW. Association of noncigarette tobacco product use with future cigarette smoking among youth in the population assessment of tobacco and health (PATH) study, 2013-2015. *JAMA pediatrics*. 2018;172(2):181-187.

- 83. Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. *Nicotine & Tobacco Research*. 2001;3(1):7-16.
- 84. Wanger JS, Culver BH. Quality standards in pulmonary function testing: past, present, future. In: American Thoracic Society; 2016.
- 85. Spindle TR, Breland AB, Karaoghlanian NV, Shihadeh AL, Eissenberg T. Preliminary results of an examination of electronic cigarette user puff topography: the effect of a mouthpiece-based topography measurement device on plasma nicotine and subjective effects. *Nicotine & Tobacco Research*. 2014;17(2):142-149.
- 86. Perkins KA, Karelitz JL, Giedgowd GE, Conklin CA. The reliability of puff topography and subjective responses during ad lib smoking of a single cigarette. *Nicotine & Tobacco Research*. 2011;14(4):490494.
- 87. Tackett AP, Lechner WV, Meier E, et al. Biochemically verified smoking cessation and vaping beliefs among vape store customers. *Addiction*. 2015;110(5):868-874.
- 88. Tackett AP, Cushing CC, Suorsa KI, et al. Illness uncertainty, global psychological distress, and posttraumatic stress in pediatric cancer: a preliminary examination using a path analysis approach. *Journal of pediatric psychology.* 2015;41(3):309-318.
- 89. Meier EM, Tackett AP, Miller MB, Grant DM, Wagener TL. Which nicotine products are gateways to regular use?: First-tried tobacco and current use in college students. *American journal of preventive medicine*. 2015;48(1):S86-S93.
- 90. Gerend MA, Newcomb ME, Mustanski B. Prevalence and correlates of smoking and e-cigarette use among young men who have sex with men and transgender women. *Drug and alcohol dependence*. 2017;179:395-399.
- 91. Buchting FO, Emory KT, Kim Y, Fagan P, Vera LE, Emery S. Transgender use of cigarettes, cigars, and e-cigarettes in a national study. *American journal of preventive medicine*. 2017;53(1):e1-e7.
- 92. Johnson SE, Holder-Hayes E, Tessman GK, King BA, Alexander T, Zhao X. Tobacco Product Use Among Sexual Minority Adults: Findings From the 2012–2013 National Adult Tobacco Survey. *American Journal of Preventive Medicine*. 2016;50(4):e91-e100.
- 93. Ganz O, Johnson AL,
- 94. AM, et al. Tobacco harm perceptions and use among sexual and gender minorities: findings from a national sample of young adults in the United States. *Addictive Behaviors*. 2018;81:104-108.
- 95. Diggle P, Liang K-Y, Zeger SL. Longitudinal data analysis. *New York: Oxford University Press.* 1994;5:13.
- 96. Curran PJ, Bauer DJ. The disaggregation of within-person and between-person effects in longitudinal models of change. *Annual review of psychology.* 2011;62:583-619.
- 97. Preacher KJ, Curran PJ, Bauer DJ. Computational tools for probing interactions in multiple linear regression, multilevel modeling, and latent curve analysis. *Journal of educational and behavioral statistics*. 2006;31(4):437-448.